CLINICAL TRIAL: NCT00815529
Title: Clinical Research on the Efficacy of Acupuncture Treatment in Chronic Low Back Pain
Status: Available | Type: Expanded Access
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Korea Health Industry Development Institute (Other Government)
Responsible Party: Mi-yeon Song, KyungHee University
Other Study IDs: KyungHU
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Last update posted 2008-12-30 (Estimated); Status verified 2008-12

CONDITIONS: Chronic Low Back Pain; Acupuncture
Keywords: Acupuncture; Chronic low back pain; Qualitative study
MeSH Terms: interventions — Acupuncture Therapy

INTERVENTIONS:
Device: Acupuncture, Pak-sham needle — 25*40mm, from 10 to 15 per each person, with the death from 5 to 20 mm, for from 15 to 20 minutes.
  Other Names: Dongbang Acupuncture Inc.

SUMMARY:
This research is planned to build a basis about effect of acupuncture for chronic low back pain with economical efficacy.

It is consisted with two sub research. First,clinical research to know the effect of acupuncture for chronic low back pain will be processed with acclate, randomized, patient, outcome-assessor masking. 130 subjects would be collected and devided into two groups(Experimental and placebo). Experimental group will undergo with real acupunture treatment twice a week, for 6 weeks and acupuncture spots would be selected for each person by clinical specialist. Placebo group will undergo with Park-sham needle and same 8 acupuncture spots would be used for all subjects also twice a week, for 6 weeks. The effect will be accessed by VAS, x-ray, ODI, SF-36, EQ-5D, BDI before and the last treatments.

Second is qualitative research to make a basis through the economic evaluation and satisfaction of acupuncture treatment for chronic low back pain. 15 persons who have been treated at oriental medical hospital for chronic low back pain and 15 in experimental group and 15 in placebo group who participate the clinical research will be collected and through the personal interview, satisfaction about the treatment and economic efficacy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The person who have been undergo chronic low back pain for chief complain over 3 months.
* The person whose age is from 18 to 65.
* The person who are normal in neurology examination.
* The person whose bothersomeness for the last week before the participation of the treatment is over VAS 5.
* The person who are diagnosed as nonspecific loe back pain.

Exclusion Criteria:

* The person who have radicular pain.
* The person who are diagnosed as specific disease which cause low back pain such as metastatic cancer, vertebral fracture, spinal infection, inflammatory spondylitis.
* The person who are diagnosed as other chronic disease which could affect the result such as caediovascular disease, diabetic neurophaty, active hepatitis, fibromyalagia, rheumatic arthritis, dementia, hemorrhagic disease, epilepsy.
* The person who have had or would have spinal surgery.
* The person who have other skeletomuscular pain as chief complain.
* The person who have been treated acupuncture treatment for low back pain last 1 month.
* The person who is taking corticosteroids, narcotics, muscle relaxant,anticoagulant drug, herb-med for low back pain, or other non-propal drugs.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Mi-yeon Song, Principal Investigator — Kyunghee University
Locations (1):
- East West Neo Medical Center, Kyung-hee university, Seoul, Gangdong-Gu, South Korea

REFERENCES:
- [Derived] Lee JH, Park HJ, Lee H, Shin IH, Song MY. Acupuncture for chronic low back pain: protocol for a multicenter, randomized, sham-controlled trial. BMC Musculoskelet Disord. 2010 Jun 14;11:118. doi: 10.1186/1471-2474-11-118. PMID 20540806